CLINICAL TRIAL: NCT04339517
Title: Postoperative Identification of Tumor Cells At the Lumpectomy Site of Patients with Early Breast Cancer
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Breast PTC
Record Dates: First submitted 2020-03-06; First posted 2020-04-09 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Aspiration of seroma fluid — Fluid will be collected from the lumpectomy site of patients between one to six weeks post-surgery and tested for the presence of persistent tumor cells (PTCs).

SUMMARY:
For early breast cancer, local surgery followed by breast radiation is a standard local treatment. It has been found that the original primary tumor site, the lumpectomy site, is the commonest location of local relapse. The researchers think that such relapse occurs because of persistent tumor cells (PTCs) at the lumpectomy site even when conventional pathology reports indicate complete resection with clear margins. The researchers propose to analyze the lumpectomy fluid (seroma) of patients who are one to six weeks post-surgery for the presence or absence of tumor cells using new technology. Results of this study may help identify women who may have increased local relapse risk beyond that suggested by conventional pathology and clinical features; it may also help identify women at very low risk of local relapse who could avoid any additional treatment after local surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Women with pathologic stage I to IIB invasive mammary breast cancer.
2. Tumor size over 1 cm.
3. Patient age 50 years or younger.
4. Primary tumor non-lobular.
5. Primary tumor non-low grade or Oncotype DX score > 18.
6. Patient is six weeks or earlier post-lumpectomy.
7. Seroma is clinically palpable and symptomatic causing discomfort and/or swelling of the lumpectomy site OR re-excision of the lumpectomy site is planned.

Max Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Identification of Persistent Tumor Cells (PTCs) | Through study completion, an average of 2 years.
  5 ml (one teaspoon) of fluid from the breast surgery site will be collected using a needle and syringe. This fluid will be sent to a laboratory in London Health Sciences Centre where it will be tested for the presence of cancer cells.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Perera, M.D., Principal Investigator — Lawson Research Institute
Locations (1):
- London Regional Cancer Program; Lawson Research Institute, London, Ontario, Canada